CLINICAL TRIAL: NCT00833625
Title: FDG-PET-CT and Biomarkers to Assess Pathologic Response in Surgical Specimens of Patients With Localized Esophageal Cancer After Chemoradiation
Brief Title: FDG-PET-CT and Biomarkers in Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-0752; PAR-08-147; NCI-2012-01614 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Gastrointestinal Disease; Esophageal Cancer
Keywords: Gastrointestinal; Esophagus; Cancer of the esophagus; Biopsy; EGD; Esophagogastroduodenoscopy; PET/CT; Positive Emission Tomography/Computerized Tomography; Esophageal Cancer; Chemoradiation; Chemotherapy; Radiation Therapy
MeSH Terms: conditions — Gastrointestinal Diseases; Esophageal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/CT Scan + Biomarkers Testing (Experimental): PET/CT scan with fluorodeoxyglucose (FDG) solution by vein, scan done 10-14 days after beginning chemotherapy and radiation (chemoradiation).
  Tissue obtained at MDACC during previous biopsy and at time of post chemoradiation surgery will be used for biomarker analysis.
  Interventions: Procedure: PET/CT (FDG PET/CT); Other: Biomarker Testings

INTERVENTIONS:
Procedure: PET/CT (FDG PET/CT) — PET/CT scan with fluorodeoxyglucose (FDG) solution by vein, scan done 10-14 days after beginning chemotherapy and radiation (chemoradiation).
  Other Names: Positron emission tomography/computed tomography
Other: Biomarker Testings — Tissue obtained at MDACC during previous biopsy and at time of post chemoradiation surgery will be used for biomarker analysis.

SUMMARY:
The goal of this clinical research study is to learn if the results of a positron emission tomography/computed tomography (PET/CT) scan done 10-14 days after beginning chemotherapy and radiation (chemoradiation) can predict how a patient with cancer of the esophagus will respond to chemoradiation. Researchers also want to learn if biomarkers (substances in the body associated with cancer) found in tumor tissue can predict response to chemoradiation.

DETAILED DESCRIPTION:
You have cancer of the esophagus and you and your doctor have agreed that you will have treatment with chemoradiation to try to shrink the cancer. You will then have surgery to remove any remaining tumor.

How well cancer of the esophagus responds to chemoradiation varies from person to person. Currently, doctors cannot tell before surgery in which patients the chemoradiation will kill all of the cancer, some of the cancer, or not much of the cancer. Studying patients' PET/CT scans and tumor tissue for biomarkers may help researchers predict how an individual patient will respond to chemoradiation. This could spare future patients from having unnecessary surgery or chemoradiation treatment that is not effective.

PET and CT scans are both standard imaging tests that doctors use to find cancer in the body. The PET scan detects the signal of actively growing cancer cells in the body and the CT scan shows the location, size, and shape of the cancer. Combining these scans provides more complete information on cancer location, growth, and changes in the cancer over time.

Currently, routine testing for esophageal cancer at MD Anderson includes a PET/CT scan at the time of diagnosis and 5 or 6 weeks after chemoradiation is completed. Researchers hope that analyzing changes seen in an "early" PET/CT scan (performed between 10-14 days after starting chemoradiation) compared to the PET/CT scan taken at the time of diagnosis may predict how well the chemoradiation will work against the patient's cancer.

PET/CT Scan:

If you are found to be eligible to take part in this study, 10-14 days after you start your chemoradiation treatment you will have a PET/CT scan performed.

You will need to fast (not have anything to eat or drink except water) for 4-6 hours before the PET/CT scan. Blood (about 1 teaspoon) will be drawn to check your blood sugar level.

You will receive a small amount of fluorodeoxyglucose (FDG) solution by vein. Cancer cells use sugar at a higher rate than normal cells do. FDG is a radioactive form of glucose (sugar) commonly used during a PET scan. The FDG helps show areas in the body where there is cancer cell growth. After receiving the FDG solution, you will rest in a quiet, darkened room for 45-60 minutes before the PET/CT scan. The entire procedure should take about 3 hours.

This PET/CT scan will be compared to your routine PET/CT scan. Your doctor will tell you of the results of this PET/CT scan. However, the results will not change the planned treatment you receive, unless the scan shows that the disease has gotten worse.

Biomarkers Testing:

Researchers will collect samples of tumor tissue previously collected at MD Anderson. This tissue will be used for biomarker testing.

Length of Study:

You will be off active study once you complete the PET/CT scan.

Medical Record Information Collection and Long-Term Follow-Up:

The study staff will collect information from your medical record on tests, evaluations, and treatments you receive as part of your routine care. The study staff will continue to collect this information from your medical record as long as you are a patient at MD Anderson.

If you stop coming to MD Anderson, you will be called by the study staff every 3 months after surgery for the first year and then every 6 months after that. During this call, you will be asked about your health status. The call should take about 5 minutes.

This is an investigational study. PET/CT scans are routine tests for patients with cancer of the esophagus. The early PET/CT scan for the purpose of this study is investigational.

Up to 95 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologic documentation of adenocarcinoma or squamous carcinoma of the esophagus at M. D. Anderson Cancer Center (MDACC).
2. Patients with localized carcinoma of the esophagus who have undergone standard testing and been evaluated by the multidisciplinary team at MDACC and are considered appropriate candidates for and are willing to undergo chemoradiation therapy followed by surgery at MDACC. Radiation may be delivered as proton or photon. These patients have clinical stage II or III cancers and they are considered medically fit to undergo surgery.
3. Patient must have undergone a baseline esophagealgastroduodenoscopy (EGD) with biopsy and endoscopic ultrasonography at MDACC, with tissue available for biomarker analysis.
4. Patient must have undergone a baseline FDG-PET/CT at MDACC or an outside institution.
5. Patient must be willing to undergo a research "early" FDG-PET/CT (12 +/- 2 days from the start of chemoradiation).
6. Patient must provide written informed consent.
7. Patient must be >/= 18 years of age.

Exclusion Criteria:

1. Patient is unable or unwilling to comply with the requirements of the protocol.
2. Patient had baseline FDG-PET/CT scan maximum SUV of < 4.0.
3. Patient is not a candidate for chemoradiation followed by surgery.
4. Patients who received induction chemotherapy prior to chemoradiation therapy are excluded.
5. Patients with T1N0 or T4anyN are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pathologic Response | PET-CT at 12 + 2 days after the start of chemoradiation
  From baseline PET-CT to "early" PET-CT [12 + 2 days after the start of chemoradiation] Frequency and percentage of pathologic complete response (pathCR) and extreme chemoradiation resistance (exCRTR) patients tabulated. Exploratory graphics, such as box plots, used to illustrate distribution of PET/CT maximum SUV by pathCR (or exCRTR) status. A logistic regression model fit for pathCR (and separately, for exCRTR), with baseline and the change of maximum SUV between baseline and early chemoradiation included as covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Elimova E, Wang X, Etchebehere E, Shiozaki H, Shimodaira Y, Wadhwa R, Planjery V, Charalampakis N, Blum MA, Hofstetter W, Lee JH, Weston BR, Bhutani MS, Rogers JE, Maru D, Skinner HD, Macapinlac HA, Ajani JA. 18-fluorodeoxy-glucose positron emission computed tomography as predictive of response after chemoradiation in oesophageal cancer patients. Eur J Cancer. 2015 Nov;51(17):2545-52. doi: 10.1016/j.ejca.2015.07.044. Epub 2015 Aug 28. PMID 26321501
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org